CLINICAL TRIAL: NCT06510868
Title: Evaluating Myelodysplastic Syndrome Risks in NET Patients Planned for Peptide Radionuclide Therapy
Acronym: MDS & PRRT
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5247
Record Dates: First submitted 2024-07-12; First posted 2024-07-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples taken for DNA/RNA/Protein analysis with storage on UHN premises. Qiagen QIAamp DNA Mini Kit will be used for extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Previous PRRT: Patients who have received PRRT within the last 4 years. There are no baseline levels available for cohort A patients. Sample size: 20.
  Interventions: Diagnostic Test: Blood collection
- Planned for PRRT: Patients who are scheduled to start PRRT in the next 3 months. Pre-PRRT clonal expansion status will only be available form this cohort. These patients will provide a comprehensive record of development of CH from exposure to PRRT. Sample size: 20.
  Interventions: Radiation: Peptide receptor radionuclide therapy (PRRT); Diagnostic Test: Blood collection
- Post PRRT Diagnosed with t-MN (MDS or AML): Patients who have t-MN (MDS or AML). Sample size: 5.
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Radiation: Peptide receptor radionuclide therapy (PRRT) — Specialized type of radionuclide therapy used to treat neuroendocrine tumors.
  Groups: Planned for PRRT
Diagnostic Test: Blood collection — Patients will have approximately 5 ml of blood drawn 6,12,24,36,48, 60 months and at the time of MDS/AML diagnosis on follow up. Genomic DNA will be extracted from serum sample using the Qiagen QIAamp DNA Mini Kit. Single-molecule molecular inversion probes (smMIPs) will be used to detect mutations. Single nucleotide variants (SNVs), short insertions and deletions (indels), and mutated myeloid genes will be captured (e.g PPM1D, DNMT3A, TET2, TP53).

SUMMARY:
This is a prospective observational study which aims to identify individuals predisposed to developing myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) could improve patient outcomes in different ways. First, it will enable improved patient selection for PRRT where alternative treatment options are available. Second, understanding the final pathway and how it is modulated by PRRT could allow the design of strategies to halt this process. Third, while it is unknown whether the development of MDS and AML is a late effect of radiopharmaceuticals in general or it is confined to cancer populations or specific radioisotopes will need to be confirmed. Finally, understanding this devastating complication is expected to be the cornerstone towards advancing radiopharmaceuticals' role in the adjuvant setting.

DETAILED DESCRIPTION:
Radiopharmaceuticals is currently used for the treatment of metastatic cancer date. While radiopharmaceuticals are generally well tolerated, one of its most devastating long-term toxicities is the development of therapy related myeloid neoplasms (t-MN), an umbrella term for myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML). PRRT (Receptor Radionuclide Therapy) is a targeted radiopharmaceutical therapy (RPT) used to treat neuroendocrine tumors. RPTs use drugs to attack cancer cells while reducing harm to healthy tissue. PRRT delivers high doses of radiation to tumors in the body to destroy or slow their growth and reduce disease side effects.

While PRRT is generally well tolerated, one of its long-term side effects is the development of therapy related myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML). The identification of genetic changes that lead to the development of MDS and AML during PRRT is a growing area of research. It is now known that the genetic changes that lead to progression into AML typically occur through many years of pre-leukemic hematopoietic stem cell clonal evolution, before development of late mutations that lead to malignant disease. The short interval between exposure to PRRT and appearance of MDS and AML would suggest some patients are already at high risk of developing AML and are potentially detectable. The ability to identify individuals predisposed to developing MDS/AML could improve patient selection for PRRT and design strategies to mitigate the development of MDS/AML.

This research proposes to study the genetic changes that occur pre-PRRT and post-PRRT using blood samples obtained from a patient population at Princess Margaret Hospital. Cohort A will consist of 20 patients that have had PRRT within the past 4 years. Cohort B will consist of 20 patients planned for PRRT. Cohort C will consist of 1-5 patients post PRRT, diagnosed with t-MN.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-3
* Life expectancy > 6 months
* Informed consent and willingness to undergoing serial genetic panel CHIP testing.
* Cohort Specific criteria

  1. Cohort A: PRRT completed within 5 years of enrolment
  2. Cohort B: PRRT planned to commence within 4 months of enrolment
  3. Cohort C: diagnosis of MDS or AML following prior PRRT.

     Exclusion Criteria:
* Unwillingness to provide blood sample and follow up as per protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This research proposes to study the genetic changes that occur pre-PRRT and post-PRRT using blood samples obtained from a patient population at Princess Margaret Hospital. Cohort A will consist of 20 patients that have had PRRT within the past 4 years. Cohort B will consist of 20 patients planned for PRRT. Cohort C will consist of 1-5 patients post PRRT, diagnosed with t-MN. In other words, patients will already be receiving PRRT or have received PRRT within 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Identify individuals predisposed to developing MDS/AML to improve patient selection for PRRT where alternative treatment options are available. | 5 years
  Determining the proportion of patients who screen positive for "prodromal AML genetic panel" pre PRRT.

SECONDARY OUTCOMES:
Detection of Genetic Mutations in the Blood Post-PRRT | 5 years
  Enrolled patients will undergo serial genetic panel testing of blood samples annually for up to 5 years to detect genetic mutations.
Assessment of Variant Allele Frequencies Post-PRRT | 5 years
  Annual genetic panel testing will be conducted to determine variant allele frequencies in the blood of patients post-PRRT for up to 5 years. The frequencies of specific gene mutations (e.g., PPM1D, TET2, DNMT3A, TP53) will be measured and analyzed in relation to clinical characteristics and treatment history.
Incidence of Therapy-Related Myeloid Neoplasms (t-MN) Post-PRRT | 5 years
  The incidence of therapy-related myeloid neoplasms (MDS and AML) will be monitored in patients post-PRRT over a 5-year follow-up period. Data will include the time to t-MN development and any associated genetic mutations identified through annual blood genetic testing.
Proportion of Patients Developing MDS/AML Post-PRRT | 5 years
  Enrolled patients will undergo annual genetic panel testing for up to 5 years to determine the proportion who develop myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) after receiving PRRT. Data collected will include baseline clinical characteristics, the amount of PRRT received, prior antineoplastic therapies, and PRRT-related adverse events to help identify factors associated with the development of these conditions.
Identification of Clonal Mutations Conferring Increased Risk of MDS/AML Post-PRRT | 5 years
  Enrolled patients will undergo annual genetic panel testing for up to 5 years to identify clonal mutations associated with an increased risk of developing myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) after receiving PRRT.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada